CLINICAL TRIAL: NCT06258707
Title: Bicentric Clinical Investigation to Assess Safety and Performance of a Hydrophobic Acrylic Enhanced Monofocal Intraocular Lens.
Brief Title: Bicentric Clinical Investigation to Assess Safety and Performance of LuxBoost IOL
Acronym: LuxBoost
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cutting Edge SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE2302; 2023-A02342-43 (Registry Identifier: French BRC Identification number)
Record Dates: First submitted 2024-02-01; First posted 2024-02-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Aphakia
Keywords: Enhanced monofocal IOL
MeSH Terms: conditions — Aphakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LuxBoost Group (Experimental): the experimental group will receive the LuxBoost intraocular lens.
  Interventions: Device: LuxBoost IOL
- LuxGood group (Active Comparator): the control group will receive the LuxGood parent intraocular lens.
  Interventions: Device: LuxGood IOL

INTERVENTIONS:
Device: LuxBoost IOL — Bilateral implantation in the capsular bag to replace the cataractous human crystalline lens.
  Arms: LuxBoost Group
Device: LuxGood IOL — Bilateral implantation in the capsular bag to replace the cataractous human crystalline lens.
  Arms: LuxGood group

SUMMARY:
The study purpose is to demonstrate safety and performance of bilateral implantation of LuxBoost intraocular lenses compared with the LuxGood Monofocal lens.

DETAILED DESCRIPTION:
The study purpose is to demonstrate safety and performance after bilateral implantation of LuxBoost intraocular lenses.

The device under investigation is a hydrophobic acrylic monofocal intraocular lens (IOL) manufactured by the sponsor of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 50 or over on the day of inclusion, presenting a
* bilateral cataract for which posterior chamber IOL implantation
* has been planned.
* Fit within the available IOL diopter range.
* Have had no previous refractive surgery.
* Regular corneal astigmatism < 1 dioptre by an automatic
* keratometer (regularity measured by topographer).
* Availability, willingness, and sufficient cognitive awareness to
* comply with examination procedures.
* Ability to attend all study follow-ups.
* Signed informed consent.

Exclusion Criteria:

* Ocular surface disease potentially affecting study results
* Subjects suffering from diagnosed degenerative visual disorders
* Pre-existing ocular pathology
* Acute or chronic disease or illness that would increase risk or confound study results
* Axial lengths and keratometry such as the IOL spherical power is
* not in the range of 14 to 28 D
* Instability of keratometry or biometry measurements
* Amblyopia
* History of ocular trauma or any prior ocular surgery including refractive procedures
* Capsular or zonular abnormalities that may affect postoperative centration or tilt of the lens

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Best corrected distance visual acuity (CDVA) | 4/6 months after surgery
  To demonstrate the non-inferiority of LuxBoost IOL compared with the LuxGood monofocal control lens in terms of best corrected distance visual acuity (CDVA) by means of statistical significance.

SECONDARY OUTCOMES:
Uncorrected Distance Visual Acuity (UDVA), Uncorrected Intermediate Visual Acuity (UIVA), Distance Corrected Intermediate Visual Acuity (DCIVA), Uncorrected Near Visual Acuity (UNVA), Distance Corrected Near Visual Acuity (DCNVA) | 4/6 months after surgery
  Photopic visual acuity at far, intermediate and near distance in monocular and binocular with LuxBoost lens compared to LuxGood lens.
Defocus curve | 4/6 months after surgery
  Binocular defocus curve with the distance correction

OTHER OUTCOMES:
Patient-reported outcomes | at preoperative visit and 4/6 months after surgery
  Patient satisfaction using Catquest-9SF questionnaire : To assess if difficulties in daily life occur due to impaired sight. This questionnaire is a 9-item Rasch-scaled instrument to assess subjective perception of visual impairment after surgery [Lundström et al, 2009]. The acceptable values are > 3.00 for differentiation between low, medium, and high abilities. Rasch analysis is commonly reported as the mean of square residual (MNSQ) and z-standardized score (ZSTD).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GUALINO, Principal Investigator — Clinique Honoré Cave 82000 Montauban; Christophe CESSES, Study Director — Cutting Edge S.A.S (Sponsor)
Locations (2):
- France (2):
  - Clinique Honore Cave, Montauban
  - West Ophta, Rennes

IPD SHARING:
Plan to Share IPD: No